CLINICAL TRIAL: NCT01017328
Title: Effect of Head Rotation on Overlap and Relative Position of Internal Jugular Vein to Carotid Artery in Infants and Children: A Study of the Anatomy Using Ultrasonography
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Hae Keum Kil / Professor, Yonsei University, College of Medicine
Other Study IDs: 4-2008-0648
Record Dates: First submitted 2009-11-19; First posted 2009-11-20 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Surgery
Keywords: infants and children undergoing surgery with general anesthesia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- surgery with general anesthesia

SUMMARY:
Effect of head rotation on overlap and relative position of internal jugular vein to carotid artery in infants and children: A study of the anatomy using ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

* Paediatric patients scheduled for elective urologic surgery were enrolled on a convenience basis, irrespective of their diagnosis or whether central venous access was planned.

Exclusion Criteria:

* Infants or children with possible c-spine disorders or haemodynamic instabilities.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: infants and children undergoing surgery with general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2009-03; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
comparison of internal jugular vein's relative position to carotid artery in children | noninvasive ultrasonographic observation after inducing general anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Hae Keum Kil, PH.D, Principal Investigator — Professor of Anesthesiology, Severance Hospital
Locations (1):
- Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea